CLINICAL TRIAL: NCT00965978
Title: A Study to Evaluate Food Effect on Pharmacokinetics Parameters After Administration of ONO-5920/YM529 Intermittent Formulation
Brief Title: A Study to Evaluate Food Effect on ONO-5920/YM529 Intermittent Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 529-CL-027
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases
Keywords: ONO-5920; YM529; Minodronic Acid; Food Effect
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases | interventions — YM 529

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose group (Experimental): Receives low dose of ONO-5920/YM529 with and without food
  Interventions: Drug: ONO-5920 / YM529
- High dose group (Experimental): Receives high dose of ONO-5920/YM529 with and without food
  Interventions: Drug: ONO-5920 / YM529

INTERVENTIONS:
Drug: ONO-5920 / YM529 — oral
  Other Names: Minodronic Acid

SUMMARY:
The aim of the study is to evaluate the effects of food intake on the plasma concentration profile of YNO-5920/YM529 in post menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women (at least 2 years after menopause)
* Body weight: more than 40.0 Kg and less than 70.0 Kg
* BMI: more than 17.6 and less than 30.0

Exclusion Criteria:

* Receives investigational drug within 120 day before the study
* Blood donation before the study
* With abnormal laboratory values

Ages: 45 Years to 81 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ONO-5920/YM529 | For 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan